CLINICAL TRIAL: NCT02980926
Title: Mepivacaine vs. Bupivacaine Spinal Anesthetic in Total Knee Arthroplasty, a Randomized Controlled Clinical Trial
Brief Title: Mepivacaine vs. Bupivacaine Spinal Anesthetic in Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, M. Chad Mahan, M.D., PGY-3, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #10455
Record Dates: First submitted 2016-09-21; First posted 2016-12-02 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Anesthesia, Spinal; Arthroplasty, Replacement, Knee; Pain Management; Early Ambulation; Ambulatory Surgical Procedures
MeSH Terms: conditions — Agnosia | interventions — Mepivacaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mepivacaine Spinal Anesthetic (Experimental): Mepivacaine 3 mL intrathecal injection of 2% solution
  Interventions: Drug: Mepivacaine
- Bupivacaine Spinal Anesthetic (Active Comparator): Bupivacaine 12 mg of 8.25% solution
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Mepivacaine — This is a shorter acting spinal anesthetic as compared to the current standard of care at this institution.
  Other Names: CAS Number: 96-88-8; Carbocaine
  Arms: Mepivacaine Spinal Anesthetic
Drug: Bupivacaine — This is the current standard of care at this institution and many centers. This is a longer acting spinal anesthetic compared to the study drug.
  Other Names: Sensorcaine; Marcaine; CAS 38396-39-3
  Arms: Bupivacaine Spinal Anesthetic

SUMMARY:
The purpose of this study is to determine if a shorter-acting spinal anesthetic called mepivacaine has advantages over a longer-acting medication called bupivacaine.

DETAILED DESCRIPTION:
Different medications last for different amounts of time and can be changed depending on the length of the procedure. A short acting spinal is generally used for procedures lasting less than 90 minutes. A longer acting medication would be any that lasts longer than 90 minutes. These medications not only block the signals that travel along the pain nerves, they also prevent the signals that tell the patients muscles to move. This means that after a total knee replacement a patient may delayed in their ability to get up and start walking early after surgery. Walking early in the recovery has been shown to decrease the rate of pulmonary embolism and death. Ambulating early is also important to prevent loss of strength, constipation, pneumonia and urinary retention.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing primary total knee arthroplasty

Exclusion Criteria:

* Chronic opioid users
* Unable to give informed consent
* Forego the use of a foley catheter
* Those with hypersensitively to amide local anesthetics or opioids
* Those with contraindications to spinal anesthesia
* Conversion to general anesthesia will be excluded.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Return of motor and sensory function | Exams will take place in 15 minute intervals beginning with arrival to the PACU and will be continued for a maximum of 6 hours or until the exam returns to baseline for 2 consecutive exams.
  Times will be recorded in minutes from the administration of the spinal anesthetic. Normal exam will include intact sensation to light touch of the thigh, calf, foot and toes. Normal motor is defined as ability to perform a straight leg raise, active knee flexion, as well as wiggling of the ankle and toes.

SECONDARY OUTCOMES:
Pain | Entire hospital admission. No data will be recorded after 96 hours.
  visual analog scale from 0 - 10
Pain | Hospital admission, maximum of 96 hours.
  morphine equivalent consumption
Time to urination | 24 hours maximum from time of spinal.
  The total time between the administration of spinal anesthesia to the first episode of spontaneous urination will be recorded. Patients who require greater than 6 hours to urinate independently are followed per hospital protocol with serial bladder scans and straight catheterization for urinary retention as needed. Patients who exceed 6 hours to urinate will be defined as having urinary retention.
Urinary retention | Entire hospital stay beginning immediately in the post operative period until discharge to a maximum of 96 hours.
  The number of straight catheterization and foley placements will be recorded as well.
Length of stay | Hospital admission maximum of 96 hours.
  Length of stay
Time to discharge readiness. | Hospital admission maximum of 96 hours.
  Time from admission to discharge readiness as assessed by physical therapy.
Transient Neurologic Symptoms | Hospital admission and first follow up visit. Data will not be recorded after 3 weeks from time of spinal
  Any episodes of transient radiating pain in the buttocks and thigh will be recorded in the hospital charts during routine post operative rounds. This is also be discussed at the first follow up visit scheduled 2 weeks after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Davis, MD, Principal Investigator — Surgeon
Locations (1):
- Henry Ford West Bloomfield, West Bloomfield, Michigan, United States

IPD SHARING:
Plan to Share IPD: No